CLINICAL TRIAL: NCT00909363
Title: Effects Of Eltrombopag On Thrombocytopenia, Platelet Function and Bleeding In Patients With Wiskott-Aldrich Syndrome/X-Linked Thrombocytopenia.
Brief Title: Thrombocytopenia and Bleeding in Wiskott-Aldrich Syndrome (WAS) Patients
Acronym: WAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: retirement of PI
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0801009600
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Wiskott-Aldrich Syndrome; Thrombocytopenia; Bleeding
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Thrombocytopenia; Hemorrhage | interventions — eltrombopag; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 1. group of 11 WAS patients treated with eltrombopag
  2. WAS patients who had their blood drawn once but did not receive eltrombopag treatment
  3. healthy children as controls for testing only
  3) healthy volunteers who had their blood drawn once
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WAS patients receiving Promacta (Experimental): Promacta® is commercially available in 12.5 mg, 25 mg, 50 mg, and 75 mg tablets. For this study, for young children unable to swallow a tablet, eltrombopag powder for oral suspension (Eltrombopag PfOS) will be used. PfOS is only available for investigational use at 20mg. Each sachet contains eltrombopag equivalent to 20mg per gm of powder and is reconstituted to a total of 10 ml so that the concentration is 2 mg/ml.
  Interventions: Drug: Promacta
- WAS patients for blood drawing only (Experimental): WAS patients not receiving treatment to serve as subjects for platelet parameter studies blood drawing once only
  Interventions: Diagnostic Test: blood drawing in patients with WAS
- healthy children for blood drawing only (Placebo Comparator): healthy children having blood obtained once as controls for platelet parameters study
  Interventions: Diagnostic Test: blood drawing in healthy controls

INTERVENTIONS:
Drug: Promacta — WAS Patients receiving treatment will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP as well as on liver tests.
  they will also have diagnostic blood testing prior to initiating treatment
  Other Names: eltrombopag, revolade
  Arms: WAS patients receiving Promacta
Diagnostic Test: blood drawing in patients with WAS — blood will be drawn for platelet parameters in WAS patients not receiving treatment either because they declined or because they were ineligible
  Arms: WAS patients for blood drawing only
Diagnostic Test: blood drawing in healthy controls — blood will be drawn once in healthy children as controls for platelet parameters
  Arms: healthy children for blood drawing only

SUMMARY:
The purpose of this project is to describe the pathophysiology of thrombocytopenia and bleeding in patients with Wiskott-Aldrich Syndrome (WAS) and determine the response to thrombopoietic agents in vitro and in vivo.

DETAILED DESCRIPTION:
Wiskott Aldrich Syndrome is an X-linked disease characterized by immunodeficiency, eczema and thrombocytopenia; a milder form of the disease known as X-Linked thrombocytopenia also exists. The thrombocytopenia in both WAS and XLT is characterized by: severe thrombocytopenia with platelet counts frequently less than 10-30,000/ul; small platelets which may be dysfunctional; and, as a result, a high rate of serious bleeding including intracranial hemorrhage.

Because eltrombopag has been shown to be remarkably efficacious in substantially increasing platelet counts in a high percentage of ITP patients, this study seeks to effectively treat patients who exhibit similar pathologies, as well as evaluate the state of platelets in patients with WAS and relate it to clinical bleeding. It also aims to demonstrate whether eltrombopag administered daily will enhance stem cell function, increase platelet production and platelet count, and reduce bleeding in patients with WAS.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for study entry, subjects must comply with the following:

* Males from 3 months old to 80 years old
* Signed written informed consent obtained prior to study entry
* Clinical diagnosis of WAS or XLT
* Platelet levels less than 100 x 109/L
* Adequate renal and hepatic function (creatinine and bilirubin less than or equal to 1.5 x IULN, AST and ALT less than or equal to 2.5 x IULN)

Exclusion Criteria:

Any patient is ineligible for study entry if he/she:

* Over the age of 80
* Women (only males are eligible)
* fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study or until at least 6 months after treatment
* Aspirin, aspirin-containing compounds, salicylates, non-steroidal anti-inflammatory medications (NSAIDS), clopidogrel or ticlopidine, warfarin or other vitamin K antagonists, unfractionated or low molecular heparin within 7 days of first infusion
* Red blood cell transfusion in the past four weeks
* Elevated (> 1.5 x ULN) prothrombin time (PT) or partial thromboplastin time (PTT)
* New York Heart Classification III or IV heart disease. Other severe cardiovascular or cardiopulmonary disease, including COPD.
* Known HIV infection, hepatitis B or C infection
* Any infection requiring antibiotic treatment within 3 days
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Prior malignancy with less than a 5-year disease-free interval, excluding nonmelanoma skin cancers and carcinoma in situ of the cervix

Ages: 3 Months to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2017-05-15 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerrits AJ, Leven EA, Frelinger AL 3rd, Brigstocke SL, Berny-Lang MA, Mitchell WB, Revel-Vilk S, Tamary H, Carmichael SL, Barnard MR, Michelson AD, Bussel JB. Effects of eltrombopag on platelet count and platelet activation in Wiskott-Aldrich syndrome/X-linked thrombocytopenia. Blood. 2015 Sep 10;126(11):1367-78. doi: 10.1182/blood-2014-09-602573. Epub 2015 Jul 29. PMID 26224646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients' families signed consents
  11 WAS patients for treatment: 1 mother signed consent but never consented to have her very young baby start study treatment (dietary issues) + 1 withdrew
  8 WAS patients' parents only were willing to have study bloods drawn
  5 normal healthy children had their parents give consent for a blood draw
Groups:
- WAS Patients Treated With Promacta: Promacta® is commercially available in 12.5 mg, 25 mg, 50 mg, and 75 mg tablets. For this study, for young children unable to swallow a tablet, eltrombopag powder for oral suspension (Eltrombopag PfOS) will be used. PfOS is only available for investigational use at 20mg. Each sachet contains eltrombopag equivalent to 20mg per gm of powder and is reconstituted to a total of 10 ml so that the concentration is 2 mg/ml.
  Promacta (eltrombopag): WAS Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
  Eltrombopag/promacta: Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
- WAS Patients for Blood Drawing Only: patients with WAS whose parents did not want them to receive treatment but were willing to let them have their blood drawn to increase the number of patients studied for platelet parameters with WAS
- Healthy Children: platelet parameters (primarily function) needed normal controls in children-----three were pre-op and two siblings were being tested as potential bone marrow donors
Period: Overall Study
Arm/Group | WAS Patients Treated With Promacta | WAS Patients for Blood Drawing Only | Healthy Children
Started | 11 | 8 | 5
Completed | 9 (1 patient started bleeding 3 days after starting eltrombopag; he underwent bone marrow transplant) | 8 | 5
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Promacta: Promacta® is commercially available in 12.5 mg, 25 mg, 50 mg, and 75 mg tablets. For this study, for young children unable to swallow a tablet, eltrombopag powder for oral suspension (Eltrombopag PfOS) will be used. PfOS is only available for investigational use at 20mg. Each sachet contains eltrombopag equivalent to 20mg per gm of powder and is reconstituted to a total of 10 ml so that the concentration is 2 mg/ml.
  Promacta (eltrombopag): Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
  Eltrombopag/promacta: Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
- Healthy Volunteers: 5 well children having blood drawn for another reason: 3 pre-op and 2 for HLAA-typing
- WAS Patients for Blood Drawing Only: patients with WAS either not eligible or not interested in eltrombpopag treatment who are willing to have their blood drawn once
- Total: Total of all reporting groups
Arm/Group | Promacta | Healthy Volunteers | WAS Patients for Blood Drawing Only | Total
Number analyzed (Participants) | 11 | 5 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 5 | 8 | 23
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 11 | 3 | 8 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 5 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: How Many WAS Patients Will Achieve Platelet Counts Above 50,000/ul.
Description: number of WAS patients achieving this increase to > 50,000/uL without rescue medication in the previous 3 weeks during eltrombopag treatment
Time Frame: 12 weeks
Population: 1 WAS subject withdrew prior to starting treatment and was not included in the analysis.
  Healthy volunteers were neither WAS patients nor received eltrombopag (both required for achievement of primary outcome #1). The WAS patients who were blood draw only also were 0 since they did not receive eltrombopag.
Measure: Number; unit: participants
Groups:
- Promacta: Promacta® is commercially available in 12.5 mg, 25 mg, 50 mg, and 75 mg tablets. For this study, for young children unable to swallow a tablet, eltrombopag powder for oral suspension (Eltrombopag PfOS) will be used. PfOS is only available for investigational use at 20mg. Each sachet contains eltrombopag equivalent to 20mg per gm of powder and is reconstituted to a total of 10 ml so that the concentration is 2 mg/ml.
  Promacta (eltrombopag): WAS Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
  Eltrombopag/promacta: Patients will start on 1 mg/kg of eltrombopag daily and be seen weekly for 12 weeks. Dose adjustment will be based on the weekly monitoring of the platelet count as utilized in ongoing studies in ITP.
- Healthy Volunteers: 8 normal subjects will be studied for degree of platelet activation from one blood draw by collaborator Alan Michelson at Boston Childrens Hospital
- Was Patients Blood Drawing Only: WAS pts who were ineligible for or did not want eltrombopag treatment
Arm/Group | Promacta | Healthy Volunteers | Was Patients Blood Drawing Only
Number analyzed (Participants) | 10 | 0 | 0
participants | 8 |  |

2. Secondary Outcome: Number of Patients With Wiskott-Aldrich Syndrome (WAS) With Grade 3 or Higher Bleeding or SAE (on WHO Scale)
Description: number of patients with bleeding SAEs while on treatment and/or number of patients with grade 3 or higher bleeding on WHO (World Health Organization) scale: the scale is from 1 to 5 with 5 = fatality and 1=very little bleeding
Time Frame: 12 Weeks
Population: 1 subject withdrew prior to starting treatment and was not included in the analysis
Measure: Number; unit: participants
Groups:
- WAS Pts: Blood Drawing Only: WASpatients who were not eligible for or did not want treatment with eltrombopag and had blood drawn once
Arm/Group | Promacta | Healthy Volunteers | WAS Pts: Blood Drawing Only
Number analyzed (Participants) | 10 | 5 | 8
participants | 1 | 0 | 0

3. Secondary Outcome: How Many Patients With WAS Had Abnormal Platelet Function Including Activation
Description: in how many patients with WAS were platelets dysfunctional or activated before treatment as measured by flow cytometry to a substantial degree and the same after treatment with eltrombopag
Time Frame: 12 weeks
Population: 1 subject withdrew prior to starting treatment and was not included in the analysis
Measure: Number; unit: participants
Groups:
- WAS Pts: Blood Drawing Only: WAS patients who are either no eligible for treatment or do not want it and agreed to have blood drawn once
Arm/Group | Promacta | Healthy Volunteers | WAS Pts: Blood Drawing Only
Number analyzed (Participants) | 10 | 5 | 8
participants | 0 | 0 | 0

4. Secondary Outcome: How Many Patients With WAS Had Substantially Increased Platelet Production After Eltrombopag
Description: in how many patients with WAS did eltrombopag increase platelet production as measured by the immature platelet fraction (IPF), a variable derived from the Sysmex auto analyzer, which is considered to be a measure of newly formed platelets ie reticulated platelets
Time Frame: 12 weeks
Population: 1 subject withdrew prior to starting treatment and was not included in the analysis. no treatment with eltrombopag was given to healthy volunteers and WAS patients who were blood drawing only so the effect of treatment in these 2 groups could not be assessed
Measure: Count of Participants; unit: Participants
Groups:
- Was Patients Blood Drawing Only: Was patients ineligible for or not interested in eltrombopag treatment
Arm/Group | Promacta | Healthy Volunteers | Was Patients Blood Drawing Only
Number analyzed (Participants) | 10 | 0 | 0
Participants | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks of treatment was the focus-----subsequent information (after 12 weeks) did not demonstrate any problems
Description: in how many patients and in how many events was there an increase in transaminases to > 2 times the upper limit of normal.
  Note, one patient was never treated and thus 10, not 11, patients were evaluable for adverse events
Groups:
- WAS Patients for Blood Drawing Only: WAS patients who are either ineligible or do not want treatment but are willing to have their blood drawn once for testing
Arm/Group | Promacta | Healthy Volunteers | WAS Patients for Blood Drawing Only
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 2/10 | 0/5 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promacta (N=10) | Healthy Volunteers (N=5) | WAS Patients for Blood Drawing Only (N=8)
bleeding SAE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — grade 3 or higher bleeding on WHO scale
increased liver tests (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) — increase in transaminases to > 2X upper limit of normal
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promacta (N=10) | Healthy Volunteers (N=5) | WAS Patients for Blood Drawing Only (N=8)
increased liver tests (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0) — transaminases > upper limit of normal but less than 2x upper limit of normal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT00909363/Prot_SAP_000.pdf